CLINICAL TRIAL: NCT01856140
Title: Treatment of Tendon Injury Using Allogenic Adipose-derived Mesenchymal Stem Cells(ALLO-ASC):A Pilot Study
Brief Title: Treatment of Tendon Injury Using Mesenchymal Stem Cells
Acronym: ALLO-ASC
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Medical Research Collaborating Center, Seoul, Korea (Other)
Responsible Party: Principal Investigator, Sun Gun Chung, Professor, Seoul National University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SNUH-RM-SGChung-ASC-01
Record Dates: First submitted 2013-04-26; First posted 2013-05-17 (Estimated); Results first posted 2022-02-18 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-02

CONDITIONS: Lateral Epicondylitis
Keywords: adipose derived mesenchymal stem cell; allogeneic stem cell
MeSH Terms: conditions — Tennis Elbow | interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 million cells/ml of ALLO-ASC (Experimental): 1 million cells/ml of ALLO-ASC(allogeneic adipose derived mesenchymal stem cell) will be injected by ultrasound guided intervention.
  Interventions: Biological: ALLO-ASC(allogeneic adipose derived mesenchymal stem cell) injection
- 10 million cells/ml of ALLO-ASC (Active Comparator): 10 million cells/ml of ALLO-ASC(allogeneic adipose derived mesenchymal stem cell) will be injected by ultrasound guided intervention.
  Interventions: Biological: ALLO-ASC(allogeneic adipose derived mesenchymal stem cell) injection

INTERVENTIONS:
Biological: ALLO-ASC(allogeneic adipose derived mesenchymal stem cell) injection

SUMMARY:
Main purpose of this study is to evaluate efficacy and safety of allogenic adipose-derived mesenchymal stem cells(ALLO-ASC) in treatment of tendon injury. ALLO-ASC will be administrated to the patients with lateral epicondylitis by ultrasonographic guided injection.

DETAILED DESCRIPTION:
Injection volume depends on the size of lesion on ultrasound examination. And all injection will be done under ultrasound guidance. First the investigators will administrate 1 million cells/ml (Group 1 for 6 participants). After monitoring the safety of injection for 2 weeks (the investigators will use WHO recommendations for grading of acute and subacute toxic effects), the investigators decide to increase the quantity as 10 million cells/ml (Group 2 for participants).

The investigators will compare the efficacy difference as quantity increase. For efficacy measurement, VAS/modified Mayo clinic performance index for elbow/lesion measurement by ultrasound will be used at 6 and 12 weeks after injections.

ELIGIBILITY:
Inclusion Criteria:

* clinically diagnosed as lateral epicondylitis (tennis elbow)
* recurrent pain in spite of conservative treatment such as physical therapy, medication, steroid injection
* symptom duration is over 6 months
* defect in common extensor tendon can be observed under ultrasound
* patient that can understand the clinical trials

Exclusion Criteria:

* patient that underwent other injection treatment within 6 weeks
* some associated diseases (such as arthritis, synovitis, entrapment of related nerve, radiculopathy to the target lesion, generalized pain syndrome, rheumatoid arthritis, pregnancy, impaired sensibility, paralysis, history of allergic or hypersensitive reaction to bovine-derived proteins or fibrin glue)
* patient that enrolled other clinical trials within 30 days
* history of drug/alcohol addiction, habitual smoker

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2018-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sun Gun Chung, MD, PhD, Principal Investigator — Seoul National University College of Medicine
Locations (1):
- Seoul National University College of Medicine, Seoul, South Korea

REFERENCES:
- [Background] Coombes BK, Bisset L, Vicenzino B. Efficacy and safety of corticosteroid injections and other injections for management of tendinopathy: a systematic review of randomised controlled trials. Lancet. 2010 Nov 20;376(9754):1751-67. doi: 10.1016/S0140-6736(10)61160-9. Epub 2010 Oct 21. PMID 20970844
- [Background] Price R, Sinclair H, Heinrich I, Gibson T. Local injection treatment of tennis elbow--hydrocortisone, triamcinolone and lignocaine compared. Br J Rheumatol. 1991 Feb;30(1):39-44. doi: 10.1093/rheumatology/30.1.39. PMID 1991216
- [Background] Sanchez M, Azofra J, Anitua E, Andia I, Padilla S, Santisteban J, Mujika I. Plasma rich in growth factors to treat an articular cartilage avulsion: a case report. Med Sci Sports Exerc. 2003 Oct;35(10):1648-52. doi: 10.1249/01.MSS.0000089344.44434.50. PMID 14523300
- [Background] Johnson GW, Cadwallader K, Scheffel SB, Epperly TD. Treatment of lateral epicondylitis. Am Fam Physician. 2007 Sep 15;76(6):843-8. PMID 17910298
- [Background] Solveborn SA, Buch F, Mallmin H, Adalberth G. Cortisone injection with anesthetic additives for radial epicondylalgia (tennis elbow). Clin Orthop Relat Res. 1995 Jul;(316):99-105. PMID 7634730
- [Background] Maffulli N, Longo UG, Denaro V. Novel approaches for the management of tendinopathy. J Bone Joint Surg Am. 2010 Nov 3;92(15):2604-13. doi: 10.2106/JBJS.I.01744. PMID 21048180
- [Background] Mishra A, Pavelko T. Treatment of chronic elbow tendinosis with buffered platelet-rich plasma. Am J Sports Med. 2006 Nov;34(11):1774-8. doi: 10.1177/0363546506288850. Epub 2006 May 30. PMID 16735582
- [Background] Kon E, Filardo G, Delcogliano M, Presti ML, Russo A, Bondi A, Di Martino A, Cenacchi A, Fornasari PM, Marcacci M. Platelet-rich plasma: new clinical application: a pilot study for treatment of jumper's knee. Injury. 2009 Jun;40(6):598-603. doi: 10.1016/j.injury.2008.11.026. Epub 2009 Apr 19. PMID 19380129
- [Background] Sanchez M, Anitua E, Azofra J, Andia I, Padilla S, Mujika I. Comparison of surgically repaired Achilles tendon tears using platelet-rich fibrin matrices. Am J Sports Med. 2007 Feb;35(2):245-51. doi: 10.1177/0363546506294078. Epub 2006 Nov 12. PMID 17099241
- [Background] Slater M, Patava J, Kingham K, Mason RS. Involvement of platelets in stimulating osteogenic activity. J Orthop Res. 1995 Sep;13(5):655-63. doi: 10.1002/jor.1100130504. PMID 7472743

RESULTS

PARTICIPANT FLOW:
Groups:
- 1 Million Cells/ml of ALLO-ASC: 1 million cells/ml of ALLO-ASC(allogeneic adipose derived mesenchymal stem cell) will be injected by ultrasound guided intervention.
  ALLO-ASC(allogeneic adipose derived mesenchymal stem cell) injection
- 10 Million Cells/ml of ALLO-ASC: 10 million cells/ml of ALLO-ASC(allogeneic adipose derived mesenchymal stem cell) will be injected by ultrasound guided intervention.
  ALLO-ASC(allogeneic adipose derived mesenchymal stem cell) injection
Period: Overall Study
Arm/Group | 1 Million Cells/ml of ALLO-ASC | 10 Million Cells/ml of ALLO-ASC
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1 Million Cells/ml of ALLO-ASC | 10 Million Cells/ml of ALLO-ASC | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 12
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.2 (8.3) | 50.5 (11.1) | 51.7 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  South Korea | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Visual Analog Scale (VAS) at 6 and 12 Weeks
Description: Self reported pain intensity during activity will be evaluated by visual analogue scale (0 = no pain, 10 = pain as bad as can be), higher scores meaning worse outcome.
Time Frame: Baseline, 6 weeks, 12 weeks after intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 1 Million Cells/ml of ALLO-ASC | 10 Million Cells/ml of ALLO-ASC
Number analyzed (Participants) | 6 | 6
score on a scale
  Baseline | 3.57 (2.1) | 3.02 (1.34)
  Post-injection 6 weeks | 2.93 (3.06) | 1.60 (1.80)
  Post-injection 12 weeks | 1.68 (1.90) | 0.87 (0.67)
Statistical Analysis 1: Comparison: 1 Million Cells/ml of ALLO-ASC vs 10 Million Cells/ml of ALLO-ASC; Null hypothesis: There is no difference between the two groups at baseline; Test type: Other; p = 0.52, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: 1 Million Cells/ml of ALLO-ASC vs 10 Million Cells/ml of ALLO-ASC; Null hypothesis: There is no difference between the two groups at post-injection 6 weeks; Test type: Other; p = 0.47, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: 1 Million Cells/ml of ALLO-ASC vs 10 Million Cells/ml of ALLO-ASC; Null hypothesis: There is no difference between the two groups at post-injection 12 weeks; Test type: Other; p = 0.52, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Modified Mayo Clinic Performance Index for the Elbow
Description: The Modified Mayo clinic performance index for the elbow measures pain, motion, stability, and daily functions. (0 to 100) Higher score means better function.
Time Frame: Baseline, 6 weeks, 12 weeks after the intervention
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | 1 Million Cells/ml of ALLO-ASC | 10 Million Cells/ml of ALLO-ASC
Number analyzed (Participants) | 6 | 6
score on a scale
  Baseline | 57.92 (15.03) | 70.00 (9.22)
  Post-injection 6 weeks | 83.75 (14.90) | 90.41 (6.97)
  Post-injection 12 weeks | 87.92 (9.41) | 91.67 (1.44)
Statistical Analysis 1: Comparison: 1 Million Cells/ml of ALLO-ASC vs 10 Million Cells/ml of ALLO-ASC; Null hypothesis: There is no difference between the two groups at baseline; Test type: Other; p = 0.227, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: 1 Million Cells/ml of ALLO-ASC vs 10 Million Cells/ml of ALLO-ASC; Null hypothesis: There is no difference between the two groups at post-injection 6 weeks; Test type: Other; p = 0.573, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: 1 Million Cells/ml of ALLO-ASC vs 10 Million Cells/ml of ALLO-ASC; Test type: Other; p = 0.588, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Defect Area of Tendon by Ultrasonography in Long Axis
Description: Defect areas were measured as the largest defect of the common extensor tendon. Higher value means larger defect area.
  With the patient supine position with the elbow in 30' flexion and full pronation, the cephalic end of the ultrasound transducer was placed on the lateral epicondyle and the long axis of the transducer was aligned with the long axis of radius. The alignment of the transducer and radius was achieved by visualizing contours of the bony structures. Multiple cross-sectional images were saved by shifting the transducer medio-laterally by 2mm at a time. Acquiring images were repeated three times.
  Among the saved images, one image showing the largest defect were selected for every patients at every time points. Manual measurements of the defect area were conducted by tracking the perimeter using ImageJ 1.48 software (National Institutes of Health, http://imagej.nih.gov/ij/) and were repeated three times by two examiners in random orders and then, averaged.
Time Frame: Baseline, 6 weeks, and 12 weeks after the intervention
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | 1 Million Cells/ml of ALLO-ASC | 10 Million Cells/ml of ALLO-ASC
Number analyzed (Participants) | 6 | 6
mm^2
  Baseline | 4197 (2607) | 5246 (2159)
  Post-injection 6weeks | 4163 (1751) | 4383 (1558)
  Post-injection 12 weeks | 2381 (1342) | 2516 (1989)
Statistical Analysis 1: Comparison: 1 Million Cells/ml of ALLO-ASC vs 10 Million Cells/ml of ALLO-ASC; Null hypothesis: There is no difference between the two groups at baseline; Test type: Other; p = 0.262, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: 1 Million Cells/ml of ALLO-ASC vs 10 Million Cells/ml of ALLO-ASC; Null hypothesis: There is no difference between the two groups at post-injection 6 weeks; Test type: Other; p = 0.631, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: 1 Million Cells/ml of ALLO-ASC vs 10 Million Cells/ml of ALLO-ASC; Null hypothesis: There is no difference between the two groups at post-injection 12 weeks; Test type: Other; p = 0.796, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Defect Area of Tendon by Ultrasonography in Short Axis
Description: Defect areas were measured as the largest defect of the common extensor tendon. Higher value means larger defect area.
  With the patient supine position with the elbow in 30' flexion and full pronation, the transducer was placed on the proximal forearm just distal to the radial head, aligning the long axis of the transducer perpendicular to the long axis of the forearm. Viewing the round radius at the horizontal center, the transducer was shifted proximally by 2mm and multiple images were saved after the transducer passed the radial head until it slid over the prominence. Acquiring images were repeated three times.
  Among the saved images, one image showing the largest defect were selected for every patients at every time points. Manual measurements of the defect area were conducted by tracking the perimeter using ImageJ 1.48 software (National Institutes of Health, http://imagej.nih.gov/ij/) and were repeated three times by two examiners in random orders and then, averaged.
Time Frame: Baseline, 6 weeks, and 12 weeks after the intervention
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | 1 Million Cells/ml of ALLO-ASC | 10 Million Cells/ml of ALLO-ASC
Number analyzed (Participants) | 6 | 6
mm^2
  Baseline | 3726 (2341) | 5018 (2494)
  Post-injection 6 weeks | 3797 (1753) | 2849 (1601)
  Post-injection 12 weeks | 2703 (1418) | 2223 (599)
Statistical Analysis 1: Comparison: 1 Million Cells/ml of ALLO-ASC vs 10 Million Cells/ml of ALLO-ASC; Null hypothesis: There is no difference between the two groups at baseline; Test type: Other; p = 0.337, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: 1 Million Cells/ml of ALLO-ASC vs 10 Million Cells/ml of ALLO-ASC; Null hypothesis: There is no difference between the two groups at post-injection 6 weeks; Test type: Other; p = 0.078, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: 1 Million Cells/ml of ALLO-ASC vs 10 Million Cells/ml of ALLO-ASC; Null hypothesis: There is no difference between the two groups at post-injection 12 weeks; Test type: Other; p = 0.439, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 52 weeks
Arm/Group | 1 Million Cells/ml of ALLO-ASC | 10 Million Cells/ml of ALLO-ASC
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 3/6 | 3/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 Million Cells/ml of ALLO-ASC (N=6) | 10 Million Cells/ml of ALLO-ASC (N=6)
Swelling at injection site (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3) — Although mild swelling was seen at the injection site in six participants (three in group 1 and three in group 2) within 48 hours after injection, the regional swelling subsided spontaneously (without any treatment) within 2 weeks.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No